CLINICAL TRIAL: NCT05250700
Title: Characterisation of Objectively Measured Physical Activity and Self-reported Habitual Exercise in Healthy Adults. An Observational Trial
Brief Title: Characterisation of Objectively Measured Physical Activity and Self-reported Habitual Exercise
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Liam Beasley, Principal Investigator, University of Bath
Other Study IDs: PA_S1_LAB
Record Dates: First submitted 2022-02-01; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults (40-70yrs)

SUMMARY:
This study aims to observe participants' physical activity (PA) using a blinded multisensor physical activity monitor as they go about their typical daily physical activities across a 6-week time frame. Participants will also complete a subjective, self-reported, online form to denote structured activities undertaken.

DETAILED DESCRIPTION:
This study will observe participants' objectively measured PA and energy expenditure in a naturalistic manner. Individuals expressing interest will be invited to attend an online familiarisation meeting to assess eligibility for the study - procedures will be presented/explained in detail before participants are given a chance to question and discuss any concerns. Once aware of the requirements, participants will be asked if they wish to take part in the main trial and asked for written informed consent.

In Visit 1 (Day 0) willing participants will then undergo a familiarisation of protocol components, and they will be provided with the SenseWear armband to be worn, constantly, over a 42-day period (except during water-based activities such as showering and swimming). The device does not include a display and so participants are blinded to the measurement. Participants will be instructed to continue with their normal lifestyles and not make any changes. On or around day 43, participants will be asked to return the device (Visit 2).

During visit 1 and visit 2 participants will be measured and weighed using a stadiometer and floor scale. Throughout the trial, weekly reminder emails will be distributed by the research team to all participants reminding them of the study requirements and providing them with an additional opportunity to raise concerns. Due to the data storage capacity of the devices, new monitors will be distributed and used monitors returned remotely via post at weeks 2 and 4.

Additionally, during this period of objective PA measurement, participants will be invited to note the start and end time of any 'structured exercise' - defined as any PA that is "planned, structured, repetitive and aimed at improving or maintaining physical fitness (Caspersen, Powell and Christenson 1985 cited by Simmich, Deacon and Russell 2019)". Participants will also be required to note time spent sleeping. Data from this self-report component of the trial will be used to demarcate bouts of purposeful, structured exercise as well as total self-reported waking time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 40-70.
* Available to attend Department for Health, University of Bath, Bath, UK.
* Capable of conducting typical daily task (e.g., housework, walking etc.).
* Willingness to wear a PA monitor for 24hr for a total of 42 days.

Exclusion Criteria:

* No cold/flu-like symptoms within the last month.
* Smokers.
* Known history of cardiac or circulatory dysfunction.
* Known to live with diabetes or other metabolic disorders.
* Known to live with severe visual or audio impairment.
* Known to live with epilepsy or have seizures.
* Known disabilities that impede daily physical activity.
* Known allergy to nickel.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from Bath and surrounding areas (South West, England) although participants able and willing to travel from further afield may be recruited. All participants are aged 40-70 years and healthy (non-clinical sample).
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Total energy expenditure [kilocalories per minute] | 6 weeks
  24-hour energy expenditure will be assessed via a wearable device enabling the estimation of total daily kilocalorie expenditure.
Domain specific energy expenditure [kilocalories per minute]. | 6 weeks
  24-hour energy expenditure will be assessed via a wearable device enabling the estimation of kilocalorie expenditure during sedentary (<1.5 metabolic equivalents) , light (1.5 - 3 metabolic equivalents), moderate (3-6 metabolic equivalents), vigorous (>6 metabolic equivalents) activities.

CONTACTS AND LOCATIONS:
Overall Officials: Liam Beasley, MSc, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Background] Simmich J, Deacon AJ, Russell TG. Active Video Games for Rehabilitation in Respiratory Conditions: Systematic Review and Meta-Analysis. JMIR Serious Games. 2019 Feb 25;7(1):e10116. doi: 10.2196/10116. PMID 30801256